CLINICAL TRIAL: NCT04226716
Title: The Role of Lumbar Proprioceptive Deficits, Psychosocial Factors and Inflammation in Pregnancy-related Pelvic Girdle Pain: a Follow-up Study in Multiparous Pregnant Women
Brief Title: The Role of Proprioceptive Deficits, Psychosocial Factors and Inflammation in Pregnancy-related Pelvic Girdle Pain
Acronym: PROFit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Lotte Janssens, Professor, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CME ZOL - CTU2019085
Record Dates: First submitted 2020-01-05; First posted 2020-01-13 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Pelvic Girdle Pain; Low Back Pain
Keywords: Postural control; Body perception; Psychosocial factors; Inflammation
MeSH Terms: conditions — Pelvic Girdle Pain; Low Back Pain; Inflammation | interventions — Psychology

STUDY DESIGN:
Intervention Model Description: Multiparous, pregnant women without PPGP at the time of inclusion are followed over a longer period of time. Assessments are performed during the first and third trimester of pregnancy and six weeks and six months postpartum.
  Nulliparous women without PPGP will be measured at one timepoint and their data are compared to those of the multiparous women.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiparous, pregnant women (Other): Multiparous women are followed over time and measurements are performed during the first and third pregnancy trimester, and six weeks and six months postpartum.
  Interventions: Behavioral: Assessment of postural control, body perception, psychosocial factors and inflammation
- Nulliparous women (Other): Nulliparous women are measured at one timepoint and their data are compared to the data of the multiparous women. Nulliparous women who take part in the reliability study are measured twice.
  Interventions: Behavioral: Assessment of postural control, body perception, psychosocial factors and inflammation

INTERVENTIONS:
Behavioral: Assessment of postural control, body perception, psychosocial factors and inflammation — Behavioral assessment of postural control, lumbar proprioceptive use during postural control, back-specific body perception, psychosocial factors (incl. perceived harmfulness of daily activities, pain-related fear of movement, fear-avoidance beliefs, (pregnancy-related) depression, anxiety and stress, optimism/pessimism, pain coping and coping with stressful life events) and inflammatory mediators

SUMMARY:
A large proportion of pregnant women develop pregnancy-related low back and/or pelvic girdle pain (PPGP), which often does not recover spontaneously postpartum. As a result, 10% of women with PPGP are thus crucial. However, the underlying mechanisms of PPGP are still poorly understood. The main objective of this study is to investigate whether lumbar proprioceptive deficits, a disturbed body perception at the lumbar spine, psychosocial factors (incl. pain-related fear of movement, depression, anxiety and stress) and increased serum concentrations of specific inflammatory mediators are associated with (1) a reduced postural control and (2) the development and/or persistence of PPGP in multiparous women during the first and third trimester of pregnancy, and six weeks and six months postpartum.

ELIGIBILITY:
Inclusion Criteria Multiparous Women:

* Singleton pregnancy
* Pregnant of second child or more than second child
* No current PPGP or did not have PPGP during current pregnancy
* Willing to provide written informed consent

Exclusion Criteria Multiparous Women:

* Pregnant for more than 16 weeks
* Having current PPGP or having had PPGP during the current pregnancy
* History of surgery/major trauma to spine or pelvis
* Surgery/physical trauma to the lower limbs more than two years ago and currently still experiencing symptoms such as pain, instability, or stiffness
* Surgery/physical trauma to the lower limbs less than two years ago
* Specific balance or vestibular disorders
* A medical diagnosis of a rheumatic condition or being under treatment for such a condition by a rheumatologist
* Neurological abnormalities (e.g., peripheral neuropathy)
* Uncorrected visual problems
* Acute ankle problems
* Being on absolute or relative bed rest due to pregnancy-related complications
* Having (had) a formal diagnosis of a psychiatric disorder
* Non-Dutch speaking

Inclusion Criteria Nulliparous Women:

* Age- and BMI- matched to pregnant participants
* Nulliparous
* Willing to provide written informed consent

Exclusion Criteria Nulliparous Women:

* Having low back or pelvic girdle pain at the time of inclusion or in the six months leading up to inclusion
* History of chronic low back or pelvic girdle pain
* History of surgery/major trauma to spine, pelvis and/or lower limbs,
* Specific balance or vestibular disorders
* Spinal deformities
* Rheumatic disease
* Neurological abnormalities
* Acute ankle problems
* (A history of) psychiatric disorders
* Uncorrected visual problems
* Non-Dutch speaking

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy-related low back and/or pelvic girdle pain (PPGP) during third gestational trimester (multiparous women) | Timepoint 2 (between gestational weeks 32-38)
  The presence of PPGP in the last month will be questioned. PPGP will be defined as: "self-reported pain in the lumbar area, between the twelfth rib and the gluteal fold, with or without pain between the posterior iliac crest and the gluteal fold, particularly in the vicinity of the sacroiliac joints that may radiate in the posterior thigh and could occur separately or in conjunction with pain in the symphysis pubis"
Pregnancy-related low back and/or pelvic girdle pain (PPGP) at six weeks postpartum (multiparous women) | Timepoint 3 (6 weeks postpartum)
  The presence of PPGP in the last two weeks will be questioned. PPGP will be defined as: "self-reported pain in the lumbar area, between the twelfth rib and the gluteal fold, with or without pain between the posterior iliac crest and the gluteal fold, particularly in the vicinity of the sacroiliac joints that may radiate in the posterior thigh and could occur separately or in conjunction with pain in the symphysis pubis"
Pregnancy-related low back and/or pelvic girdle pain (PPGP) at six months postpartum (multiparous women) | Timepoint 4 (6 months postpartum)
  The presence of PPGP in the last two weeks will be questioned. PPGP will be defined as: "self-reported pain in the lumbar area, between the twelfth rib and the gluteal fold, with or without pain between the posterior iliac crest and the gluteal fold, particularly in the vicinity of the sacroiliac joints that may radiate in the posterior thigh and could occur separately or in conjunction with pain in the symphysis pubis"
Postural control during first gestational trimester (multiparous women) | Timepoint 1 (before gestational week 16)
  Upright standing balance control will be measured as center-of-pressure displacements with a force plate.
Postural control during third gestational trimester (multiparous women) | Timepoint 2 (between gestational weeks 32-38)
  Upright standing balance control will be measured as center-of-pressure displacements with a force plate.
Postural control (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion), (Timepoint 2 (1 - 2 weeks after Timepoint 1))
  Upright standing balance control will be measured as center-of-pressure displacements with a force plate.

SECONDARY OUTCOMES:
Disability due to PPGP with the Modified Low Back Pain Disability Questionnaire (MDQ) (multiparous women) | Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The MDQ quantifies the extent of functional limitation in daily life due to low back pain: 10 items, total score range 0 - 100. Higher scores indicate higher levels of disability.
Disability due to low back pain with the Modified Low Back Pain Disability Questionnaire (MDQ) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The MDQ quantifies the extent of functional limitation in daily life due to low back pain: 10 items, total score range 0 - 100. Higher scores indicate higher levels of disability.
Disability due to PPGP with the Quebec Back Pain Disability Scale (QBPDS) (multiparous women) | Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The QBPDS assesses disability in individuals with low back pain and PPGP: 20 items, total score range 0 - 100. Higher scores indicate higher levels of disability.
Pain intensity of PPGP with Numerical Pain Rating Scale (NPRS) (multiparous women) | Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  Pain intensity will be rated on the NPRS that ranges from 0 ("no pain") to 10 ("the worst pain imaginable").
Pain location of PPGP with a body chart (multiparous women) | Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  Individuals with PPGP will indicate the pain locations on a body chart.
Current body weight (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  Current body weight will be measured (kg)
Current body weight (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  Current body weight will be measured (kg)
Current body composition (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  Current body composition will be measured with bioelectrical impedance analysis.
Proprioceptive use during postural control (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38)
  Center-of-pressure displacements in response to ankle muscle and lower back muscle vibration (60 Hz, 15s) during upright standing will be measured with a force plate.
Proprioceptive use during postural control (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion), Timepoint 2 (1-2 weeks after Timepoint 1)
  Center-of-pressure displacements in response to ankle muscle and lower back muscle vibration (60 Hz, 15s) during upright standing will be measured with a force plate.
Body perception at the lumbar spine will be assessed with a laterality recognition task ("Recognise Back" app) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  During the laterality recognition task, participants view 40 pictures of a model that has its lower back bent or rotated to the left or the right side. They will be asked to judge the direction of movement as quickly and accurately as possible. Average speed (in seconds) of response time and average accuracy of the answers (in %) will be recorded.
Body perception at the lumbar spine will be assessed with a laterality recognition task ("Recognise Back" app) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion), Timepoint 2 (1-2 weeks after Timepoint 1)
  During the laterality recognition task, participants view 40 pictures of a model that has its lower back bent or rotated to the left or the right side. They will be asked to judge the direction of movement as quickly and accurately as possible. Average speed (in seconds) of response time and average accuracy of the answers (in %) will be recorded.
Body perception at the lumbar spine will be assessed with the Fremantle Back Awareness Questionnaire (FreBAQ) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The FreBAQ assesses back-specific body perception: 9 items, total score range 0 - 45. Higher score indicate a more disturbed body perception.
Body perception at the lumbar spine will be assessed with the Fremantle Back Awareness Questionnaire (FreBAQ) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The FreBAQ assesses back-specific body perception: 9 items, total score range 0 - 45. Higher score indicate a more disturbed body perception.
Pain-related fear of movement with the Tampa Scale for Kinesiophobia (TSK) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The TSK evaluates fear of movement and pain-related fear: 17 items, total score range 17 - 68. Higher scores indicate higher levels of pain-related fear of movement.
Pain-related fear of movement with the Tampa Scale for Kinesiophobia (TSK) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The TSK evaluates fear of movement and pain-related fear: 17 items, total score range 17 - 68. Higher scores indicate higher levels of pain-related fear of movement.
Perceived harmfulness of specific physical activities with the Photograph Series of Daily Activities - Short Electronic Version (PhoDA-SEV) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  During the PhoDA-SEV, participants view 40 pictures of daily life activities. They will be asked to imagine themselves performing the depicted activity and to indicate to which extent they believe that the activity is harmful to their back on a scale from 0 ("not harmful at all") to 100 ("extremely harmful"): 40 items, total score range 0 - 100. Higher scores indicate a higher perceived harmfulness of physical activities.
Perceived harmfulness of specific physical activities with the Photograph Series of Daily Activities - Short Electronic Version (PhoDA-SEV) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  During the PhoDA-SEV, participants view 40 pictures of daily life activities. They will be asked to imagine themselves performing the depicted activity and to indicate to which extent they believe that the activity is harmful to their back on a scale from 0 ("not harmful at all") to 100 ("extremely harmful"): 40 items, total score range 0 - 100. Higher scores indicate a higher perceived harmfulness of physical activities.
Fear avoidance beliefs with the Fear-Avoidance Beliefs Questionnaire (FABQ) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The FABQ consists of 16 statements for which the participant rates her agreement with the statement on a scale from 0 ("completely disagree") to 6 ("completely agree"): 16 items, total score range 0 - 96). Higher scores indicate that poorer fear avoidance beliefs are held.
Fear avoidance beliefs with the Fear-Avoidance Beliefs Questionnaire (FABQ) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The FABQ consists of 16 statements for which the participant rates her agreement with the statement on a scale from 0 ("completely disagree") to 6 ("completely agree"): 16 items, total score range 0 - 96). Higher scores indicate that poorer fear avoidance beliefs are held.
Catastrophic thinking related to pain with the Pain Catastrophizing Scale (PCS) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The PCS contains 13 statements on thoughts and emotions possibly related to the experience of pain, for which the participants rates her agreement: 13 items, total score range 0 - 52. Higher scores indicate higher levels of pain catastrophizing.
Catastrophic thinking related to pain with the Pain Catastrophizing Scale (PCS) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The PCS contains 13 statements on thoughts and emotions possibly related to the experience of pain, for which the participants rates her agreement: 13 items, total score range 0 - 52. Higher scores indicate higher levels of pain catastrophizing.
Pregnancy-related depression with the Edinburgh Depression Scale (EDS) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The EDS evaluates perinatal depression: 10 items, total score range 0 - 30. Higher scores indicate higher levels of pregnancy-related depression.
Pregnancy-related anxiety with the Revised Pregnancy-related Anxiety Questionnaire (PRAQ-R2) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The PRAQ-R2 evaluates pregnancy-related anxiety: 10 items, total score range 10 - 50. Higher scores indicate higher levels of pregnancy-related anxiety.
Pregnancy-related stress with the Tilburg Pregnancy Distress Scale (TPDS) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The TPDS assesses pregnancy-related distress: 16 items, total score range 0 - 48). Higher scores indicate higher levels of pregnancy-related stress.
Depression, anxiety and stress in general with the Depression Anxiety Stress Scale (DASS-21) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The DASS-21 evaluates depressive mood, anxiety and stress in general: 21 items, total score per subscale (Depression, Stress, Anxiety) range 0 - 21. Higher scores indicate higher levels of depressive mood (DASS-21-Depression), anxiety (DASS-21-Anxiety) and stress (DASS-21-Stress).
Depression, anxiety and stress in general with the Depression Anxiety Stress Scale (DASS-21) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The DASS-21 evaluates depressive mood, anxiety and stress in general: 21 items, total score per subscale (Depression, Stress, Anxiety) range 0 - 21. Higher scores indicate higher levels of depressive mood (DASS-21-Depression), anxiety (DASS-21-Anxiety) and stress (DASS-21-Stress).
Negative and positive affect, hedonic tone and independent variables (including cognitive and overall functioning, meaningful life and happiness) with the Leuven Affect Pleasure Scale (LAPS) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The LAPS comprehensively evaluates negative and positive affect, hedonic tone and independent variables (including cognitive and overall functioning, meaningful life and happiness): 16 items. It contains three subscores, which are calculated by adding the score on items 1-4 (Negative Affect), items 5-8 (Positive Affect) and items 9-12 (Hedonic Tone). Negative Affect subscale: 4 items, score range 0 - 40, higher scores indicate higher levels of negative affect. Positive Affect subscale: 4 items, score range 0 - 40, higher scores indicate higher levels of positive affect. Hedonic Tone subscale: 3 items, total score range 0 - 30, higher scores indicate higher levels of hedonic tone.
Negative and positive affect, hedonic tone and independent variables (including cognitive and overall functioning, meaningful life and happiness) with the Leuven Affect Pleasure Scale (LAPS) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The LAPS comprehensively evaluates negative and positive affect, hedonic tone and independent variables (including cognitive and overall functioning, meaningful life and happiness): 16 items. It contains three subscores, which are calculated by adding the score on items 1-4 (Negative Affect), items 5-8 (Positive Affect) and items 9-12 (Hedonic Tone). Negative Affect subscale: 4 items, score range 0 - 40, higher scores indicate higher levels of negative affect. Positive Affect subscale: 4 items, score range 0 - 40, higher scores indicate higher levels of positive affect. Hedonic Tone subscale: 3 items, total score range 0 - 30, higher scores indicate higher levels of hedonic tone.
Generalized anxiety with the 7-item Generalized Anxiety Disorders scale (GAD-7) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The GAD-7 evaluates generalized anxiety: 7 items, total score range 0 - 21.
Generalized anxiety with the 7-item Generalized Anxiety Disorders scale (GAD-7) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The GAD-7 evaluates generalized anxiety: 7 items, total score range 0 - 21.
The emotional bond between mother and child with the Maternal Antenatal/Postpartum Attachment Scale (MAAS/MPAS). | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The MAAS evaluates the emotional bond between mother and child antenatally, while the MPAS assesses this bond postnatally: 19 items, total score range 0 - 95
Pain coping strategies with the Pain Coping Inventory (PCI) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The PCI evaluates whether one uses passive or active coping strategies: 34 items, total score range 0 - 100
Pain coping strategies with the Pain Coping Inventory (PCI) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The PCI evaluates whether one uses passive or active coping strategies: 34 items, total score range 0 - 100
Optimism and pessimism with the Life Orientation Test Revised (LOT-R) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The LOT-R contains 10 items: 3 evaluating optimism, 3 evaluating pessimism and 4 filler items, total score range on each subscale (optimism, pessimism) 0 - 12.
Optimism and pessimism with the Life Orientation Test Revised (LOT-R) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The LOT-R contains 10 items: 3 evaluating optimism, 3 evaluating pessimism and 4 filler items, total score range on each subscale (optimism, pessimism) 0 - 12.
The ability to cope in a stressful situation with the Sense of Coherence Scale (SOC-13) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The SOC-13 contains 13 items, total score ranges 0 - 91
The ability to cope in a stressful situation with the Sense of Coherence Scale (SOC-13) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The SOC-13 contains 13 items, total score ranges 0 - 91
Pain frequency of PPGP (multiparous women) | Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  Pain frequency will be assessed with the question: 'How often do you experience pain?' Response options will include: Some days (1), Most days (2), and Every day (3).
Health-related quality of life with the 36-Item Short Form Health Survey (SF-36) (multiparous women) | Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The SF-36 evaluates health-related quality of life, 8 scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Scores for the different scales are converted and pooled using a scoring key, for a total score ranging 0 - 100
Health-related quality of life with the 36-Item Short Form Health Survey (SF-36) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The SF-36 evaluates health-related quality of life, 8 scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Scores for the different scales are converted and pooled using a scoring key, for a total score ranging 0 - 100
Inflammation with blood samples (multiparous women) | Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  Serum concentrations of inflammatory mediators will be measured in a blood sample.

OTHER OUTCOMES:
Diagnostic clinical tests for PPGP (multiparous women) | Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The following pain provocation tests for PPGP will be performed: thigh thrust and trendelenburg test. A score of 1 will be assigned to each test that provokes the participants' pain, a score of 0 will be assigned to each test that does not provoke the pain. All scores will be combined into one overall score.
Ability to transfer load between the spine and the legs via the pelvis with active straight leg raise test (ASLR) (multiparous women) | Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The participant will perform the ASLR test in supine lying: she will be asked to lift one leg 20 cm off the bed, and a score between 0 and 5 will be assigned depending on the difficulty experienced (0= "not difficult at all, 1= minimally difficult, 2= somewhat difficult, 3 = fairly difficult, 4= very difficult, 5= unable to do).
Sociodemographic information: age (multiparous women) | Timepoint 1 (before gestational week 16)
  The age of the participant will be noted (in years)
Sociodemographic information: age (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The age of the participant will be noted (in years)
Sociodemographic information: annual household income (multiparous women) | Timepoint 1 (before gestational week 16)
  Annual household income will be questioned (in Euro)
Sociodemographic information: annual household income (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  Annual household income will be questioned (in Euro)
Sociodemographic information: marital status (multiparous women) | Timepoint 1 (before gestational week 16)
  Marital status be questioned (single, married/registered partnership)
Sociodemographic information: marital status (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  Marital status be questioned (single, married/registered partnership)
Sociodemographic information: educational level (multiparous women) | Timepoint 1 (before gestational week 16)
  The highest degree obtained will be recorded.
Sociodemographic information: educational level (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The highest degree obtained will be recorded.
Sociodemographic information: current profession (multiparous women) | Timepoint 1 (before gestational week 16)
  The current profession will be recorded, as well as the type of work (sedentary work, manual work, heavy work)
Sociodemographic information: current profession (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The current profession will be recorded, as well as the type of work (sedentary work, manual work, heavy work)
Number of previous pregnancies (multiparous women) | Timepoint 1 (before gestational week 16)
  The number of previous pregnancies will be recorded.
Number of previous child deliveries (multiparous women) | Timepoint 1 (before gestational week 16)
  The number of previous child deliveries will be recorded.
Number of stillbirths and live births (multiparous women) | Timepoint 1 (before gestational week 16)
  The number of stillbirths and live births will be recorded.
Number of previous miscarriages (multiparous women) | Timepoint 1 (before gestational week 16)
  The number of previous miscarriages will be recorded.
Job status (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  Job status will be recorded (i.e., working full-time, working part-time, in sick leave)
Sick Leave (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  In case of sick leave, we will ask whether this is pregnancy-related or not, and the total number of sick leave days will be noted.
Job status (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  Job status will be recorded (i.e., working full-time, working part-time, in sick leave)
Sick Leave (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  In case of sick leave, we will ask whether this is pregnancy-related or not, and the total number of sick leave days will be noted.
Tobacco use (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  Smoking habits will be questioned by using the following categories: every day smoker (smokes now and smokes every day), someday smoker (smokes now, but not every day), former smoker (has quit smoking), never smoker
Tobacco use (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  Smoking habits will be questioned by using the following categories: every day smoker (smokes now and smokes every day), someday smoker (smokes now, but not every day), former smoker (has quit smoking), never smoker
Alcohol use (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  Alcohol use will be questioned by using the following categories: every day drinker (drinks now and drinks every day), someday drinker (drinks now, but not everyday), former drinker (has quit drinking now), never drinker.
Alcohol use (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  Alcohol use will be questioned by using the following categories: every day drinker (drinks now and drinks every day), someday drinker (drinks now, but not everyday), former drinker (has quit drinking now), never drinker.
Habitual physical activity (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  Habitual physical activity will be questioned using the following categories: no physical activity, physical activity, but less than recommended (<150min moderate intensity/week), physical activity, as recommended.
Habitual physical activity (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  Habitual physical activity will be questioned using the following categories: no physical activity, physical activity but less than recommended (<150min moderate intensity/week), physical activity as recommended.
Subjective sleep quality with the Pittsburgh Sleep Quality Index (PSQI) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The PSQI assesses sleep quality over the past month: 19 items, global sleep quality scores range 0 - 21
Subjective sleep quality with the Pittsburgh Sleep Quality Index (PSQI) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  The PSQI assesses sleep quality over the past month: 19 items, global sleep quality scores range 0 - 21
Height (multiparous women) | Timepoint 1 (before gestational week 16)
  Height will be measured and reported in cm.
Height (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion)
  Height will be measured and reported in cm.
Pre-pregnancy body weight (multiparous women) | Timepoint 1 (before gestational week 16)
  Pre-pregnancy body weight will be questioned and reported in kg.
Number of falls during previous pregnancies (multiparous women) | Timepoint 1 (before gestational week 16)
  The number of falls experienced during previous pregnancies will be noted. The following question will be asked: "During your previous pregnancies, did you experience any loss of balance, resulting in a fall where some part of your body--other than your feet--touched the ground?"
Gestational week during which fall occurred during previous pregnancies (multiparous women) | Timepoint 1 (before gestational week 16)
  If the participant experienced a fall during a previous pregnancy, the gestational week during which the fall(s) occurred will be noted.
Situation during which fall occurred during previous pregnancies | Timepoint 1 (before gestational week 16)
  If the participant experienced a fall during a previous pregnancy, the situation during which the falls occurred will be noted, by using the following categories: trip, slip, during stair ascent, during stair descent, during athletic activity.
Injury severity of falls that occurred during previous pregnancies (multiparous women) | Timepoint 1 (before gestational week 16)
  If the participant experienced a fall during a previous pregnancy, the injury severity associated with the falls will be noted by using the following categories: no injury, mild injury requiring home treatment, major injury requiring medical attention
Urinary incontinence during previous pregnancies (multiparous women) | Timepoint 1 (before gestational week 16)
  The presence of urinary incontinence during previous pregnancies (yes/no), and the recovery of urinary incontinence postpartum (full, partial, no recovery) will be questioned.
Anal incontinence during previous pregnancies (multiparous women) | Timepoint 1 (before gestational week 16)
  The presence of incontinence for stool and gas during previous pregnancies (yes/no), and the recovery of incontinence for stool and gas postpartum (full, partial, no recovery) will be questioned.
Information on previous deliveries: Date of delivery (multiparous women) | Timepoint 1 (before gestational week 16)
  We will ask whether the previous children date of delivery
Information on previous deliveries: vaginal delivery or caesarean section (multiparous women) | Timepoint 1 (before gestational week 16)
  We will ask whether the previous deliveries were vaginal deliveries of caesarean sections.
Information on previous deliveries: episiotomy or vaginal tear | Timepoint 1 (before gestational week 16)
  Information on presence of episiotomy (yes/no) and occurrence of vaginal tear (yes/no) in previous deliveries will be collected.
Information on previous deliveries: Assistance of instrument during delivery (multiparous women) | Timepoint 1 (before gestational week 16)
  We will ask whether an instrument was used during the delivery: forceps, vacuum cup,...
Information on previous deliveries: Assisted reproductive treatment (multiparous women) | Timepoint 1 (before gestational week 16)
  We will ask whether the women are pregnant through assisted reproductive treatment
Number of falls during current pregnancy or in postpartum period (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  The number of falls experienced during the current pregnancy or postpartum period will be noted. The following question will be asked: "Did you experience any loss of balance, resulting in a fall where some part of your body--other than your feet--touched the ground?"
Timepoint during which fall occurred during current pregnancy or postpartum period (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  If the participant experienced a fall during or after the current pregnancy, the timepoint during which this fall occurred wil be noted.
Situation during which fall occurred during current pregnancy or postpartum period (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  If the participant experienced a fall during or after the current pregnancy, the situation during which the falls occurred will be noted, by using the following categories: trip, slip, during stair ascent, during stair descent, during athletic activity.
Injury severity of falls that occurred during current pregnancy or postpartum period (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  If the participant experienced a fall during or after the current pregnancy, the injury severity associated with the falls will be noted by using the following categories: no injury, mild injury requiring home treatment, major injury requiring medical attention
Urinary incontinence during current pregnancy (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38), Timepoint 3 (6 weeks postpartum) and Timepoint 4 (6 months postpartum)
  Urinary incontinence will be evaluated with the Pelvic Floor Distress Inventory (PFDI-20). The PFDI-20 contains 20 items, total score range 0 - 300
Information on current pregnancy: Assisted reproductive treatment (multiparous women) | Timepoint 1 (before gestational week 16)
  We will ask whether the women are pregnant through assisted reproductive treatment
Information on current pregnancy: Morning sickness | Timepoint 1 (before gestational week 16)
  We will ask whether the women experience morning sickness during their current pregnancy.
Information on child delivery: Date of delivery (multiparous women) | Timepoint 3 (6 weeks postpartum)
  We will ask the date of delivery.
Information on child delivery: episiotomy or vaginal tear (multiparous women) | Timepoint 3 (6 weeks postpartum)
  Information on presence of episiotomy (yes/no) and occurrence of vaginal tear (yes/no) will be collected
Information on child delivery: Assistance of instrument during delivery (multiparous women) | Timepoint 3 (6 weeks postpartum)
  We will ask whether an instrument was used during the delivery: forceps, vacuum cup,...
Fear of falling during postural control measurements with Numerical Rating Scale (NRS) (multiparous women) | Timepoint 1 (before gestational week 16), Timepoint 2 (between gestational weeks 32-38)
  Fear of falling during postural control measurements will be rated after each measurement on the NRS that ranges from 0 ("no fear") to 10 ("the worst fear imaginable").
Fear of falling during postural control measurements with Numerical Rating Scale (NRS) (nulliparous women) | Timepoint 1 (within 2 weeks after inclusion), (Timepoint 2 (1 - 2 weeks after Timepoint 1))
  Fear of falling during postural control measurements will be rated after each measurement on the NRS that ranges from 0 ("no fear") to 10 ("the worst fear imaginable").

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Janssens, PhD, PT, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No